CLINICAL TRIAL: NCT07149753
Title: Pilot Study: Safety and Therapeutic Dose of a Miltefosine Gel (G-MTF) in Patients With Uncomplicated Cutaneous Leishmaniasis (NCCL)
Brief Title: Pilot Study: Miltefosine Gel (G-MTF) in Patients With Cutaneous Leishmaniasis
Acronym: G-MTF01
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Universidad Industrial de Santander (Other)
Collaborators: Fundación Oftalmológica de Santander Clínica Carlos Ardila Lulle (Other)
Responsible Party: Principal Investigator, Patricia Escobar, Professor, PhD, Universidad Industrial de Santander
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1102-890-82095; Grant 2022-0645 (Other Grant/Funding Number: MinCiencias)
Record Dates: First submitted 2025-08-16; First posted 2025-09-02 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Cutaneous Leishmaniasis; Cutaneous Leishmaniasis, American; Topical Administration
Keywords: cutaneous leishmaniasis; topical treatment; miltefosine; hydrogel
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis, Mucocutaneous | interventions — miltefosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MILTEFOSINE hydrogel 0.5% (Experimental): MILTEFOSINE hydrogel 0.5% topically daily for 28 days
  Interventions: Drug: MILTEFOSINE gel
- MILTEFOSINE hydrogel 1.0% (Experimental): MILTEFOSINE hydrogel 1.0% topically daily for 28 days
  Interventions: Drug: MILTEFOSINE gel
- MILTEFOSINE hydrogel 1.5% (Experimental): MILTEFOSINE hydrogel 1.5% topically daily for 28 days
  Interventions: Drug: MILTEFOSINE gel

INTERVENTIONS:
Drug: MILTEFOSINE gel — Each patient will receive a 30 g tube of G-MTF with instructions and recommendations for use. The first dose will be in the FOSCAL clinical studies unit; subsequent doses will be applied at the patient's site of origin based on their autonomy, once a day (morning or night). Instructions include washing hands thoroughly, cleaning the lesion, applying a thin layer of gel, leaving it uncovered for at least 15 minutes, avoiding contact with water until the next dose, and storing the gel properly during treatment.
  Other Names: topical miltefosine

SUMMARY:
The goal of this clinical trial is to learn if the drug MILTEFOSINE, used topically in a hydrogel, works to treat non-complicated cutaneous leishmaniasis (CL) in adults. It will also learn about the safety of the drug MILTEFOSINE used topically. The main questions it aims to answer are:

* Is topical treatment with MILTEFOSINE hydrogel effective in patients with CL, thus justifying its continuation in the clinical phases (II and III) of development?
* What skin problems do participants have when using miltefosine hydrogels over CL lesions? Researchers will evaluate the safety and effectiveness of various concentrations of MILTEFOSINE hydrogel: 0.5%, 1.0%, and 1.5%.

Participants will:

* Apply the MILTEFOSINE hydrogel to the affected lesions daily for 28 consecutive days.
* Visit the Center at least two days prior to the study. This initial visit will include diagnostic tests, interviews, study information, informed consent, and the administration of the first doses. After this, patients are required to return to the clinic on day 28 and again three months later for additional check-ups and tests.
* Take a photo once a week for checkups, and keep a note of their symptoms

DETAILED DESCRIPTION:
Study universe/study population It is the department of Santander in Colombia. The department ranks third in Colombia for the highest number of CL cases, with an incidence of 57% of cases per 100,000 inhabitants at risk. Additionally, several endemic regions of leishmaniasis are situated near the city of Floridablanca, where the facilities of the Clinical Study Center of the Santander Ophthalmological Foundation (FOSCAL) are located, and this will be the study site. The study population includes patients with ncCL who live in endemic leishmaniasis areas within Santander. For selecting the study population, support from the Ministry of Health of Santander (SSS) will be available. The target population resides in endemic areas for CL within Santander, particularly in the municipal villages of Rionegro, Playón, Landázuri, San Vicente de Chucuri, and Cimitarra. Recruitment of patients will be conducted in three ways: face-to-face in the municipal capitals, with direct communication to residents under the guidance and supervision of the Office of Vector-Borne Diseases (ETV) of the SSS; through printed advertising, such as posters and brochures; and virtually via social networks.

Sample size This project is a pilot study, so the sample size is based on convenience. Consequently, the sample will include 15 participants (experimental group 1: n = 5; experimental group 2: n = 5; experimental group 3: n = 5). The sample size was determined considering: (i) the flow of patients in the institution (consultation estimates for this condition); (ii) the challenges in mobilising patients from endemic areas for this condition; and (iii) the resources available from the sponsoring organisation. This study will establish the clinical and statistical groundwork needed for future larger-scale studies by estimating the treatment response in the selected population.

Previus steps Patients will be informed about the study's objectives and potential risks associated with participation. A web application called "leishmaniasis-CINTROP" will be installed and demonstrated to serve as support and a permanent point of contact with us. Those wishing to participate must sign the informed, reviewed, validated, and approved consent before any intervention. The pre-treatment or screening period will last from 1 to 4 days, during which patients will be verified for inclusion criteria, and a general medical examination, electrocardiogram (ECG), blood chemistry tests (including transaminases, amylase, lipase, and creatinine), and parasitological diagnosis will also be performed. Patients meeting the requirements will be eligible to participate. A woman of reproductive age should be asked to take a pregnancy test. She must guarantee the use of an effective contraceptive method during treatment and for up to three months thereafter. The medical history of each participant will be recorded and managed in accordance with Resolution 1995 of 1999. It will consist of sections such as personal data, personal and family history, habits (physical activity, smoking, alcohol consumption, others), diagnoses (for leishmaniasis or other vector-borne diseases), physical examination (vital signs), site of injury(s), treatment assignment (code), treatment follow-up record, and adverse event reporting.

A general examination will be conducted by an internist with extensive knowledge of the study and the disease, during which data for the medical history will be recorded, including details on the progression of the injury(s). Vital signs, weight, and height will be measured. An electrocardiogram (ECG) will be performed on all patients and analysed to ensure the sinus rhythm, P wave, QRS complex, and T wave are within normal parameters.

For biochemical tests, diagnosis, and parasite culture, the following procedures will be used. A sample will be collected through venipuncture into a tube without an anticoagulant. The samples will then be centrifuged at 3500 rpm for 10 minutes. Levels of transaminases (aspartate aminotransferase [AST] and alanine aminotransferase [ALT]), amylase, lipase, and creatinine will be measured using validated methods by a laboratory certified in Good Clinical Practice (GCP). All women will be tested for pregnancy using commercial tests.

Regarding procedures for patients' injuries, the following steps will be taken: to collect imprints used in leishmaniasis diagnosis, the lesion will be carefully cleaned with gauze and a saline solution. A local anaesthetic (such as lidocaine) may be applied if necessary or recommended by the physician, approximately 20 minutes before proceeding. A sample (imprint) will be obtained by inserting the tip of a scalpel into the edge of the lesion, and the material will be spread on a glass slide. This smear will be fixed with alcohol, stained with Giemsa, and examined microscopically at 1000x magnification. The presence of at least one amastigote will be considered a positive result.

Randomisation Patients will be randomly allocated on a one-to-one basis using IVRS software "Interactive Voice/Web Response System in Clinical Research" for each treatment arm, with a code assigned for procedures and follow-up. Randomisation will be carried out in bulk, with the list prepared prior to the start of the study. The candidate who meets the inclusion and exclusion criteria will be assigned to the next available study group on the list. If a patient exits the study before treatment allocation is complete or before the therapy phase begins, their position on the list will be filled by the next candidate. Both the study investigators and the patients will be aware of their group allocation, as there will be no masking of treatments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of confirmed cutaneous leishmaniasis (CL)
* Age: 18 - 65 years.
* Patients who have 1-4 CL skin lesions with a diameter of 1-4 cm, with an evolution time of more than one month and not located on the face, ears, or joints.
* Patients WITHOUT suspected complicated CL (large regional lymphadenopathy, several large lesions spread to different parts of the body); NO mucosal leishmaniasis and NO suspicion of unusual leishmaniasis syndromes (e.g., recurrent leishmaniasis, diffuse or disseminated CL).
* Patients with NO history of systemic antileishmania treatment within 8 weeks prior to starting the study.
* Patients WITHOUT treatment failure with local therapy (intralesional antimonial injections or thermotherapy) or systemic therapy.

Exclusion Criteria:

* Pregnant or lactating women; women of reproductive age who refuse to use contraception until 45 days after treatment ends.
* Patients with cardiovascular, hepatic, or renal impairment or who report underlying diseases that medically compromise their participation in this study.
* Patients who report a history of immunodeficiency.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
End of treatment (lesion healing) | 28 days
  Percentage change in lesion size: Compared to baseline (the size before treatment).

SECONDARY OUTCOMES:
Post-treatment (lesion healing or lesion reduction) | 90 days
  Percentage change in lesion size: Compared to baseline (the size before treatment). Lesion healing:
  A patient will be considered "cure" if they achieve 100% epithelialisation of the lesion (total reduction of the lesion with the presence of scar) without relapse for up to 3 months post-treatment. Therapeutic failure is defined as an increase in the lesion area to twice its initial size at the end of treatment or if the lesion does not reduce by more than 50% at three months post-treatment. Relapse is noted if, after reducing by more than 50%, the lesion enlarges again, reaching or exceeding its original size during the three months post-treatment.
Number and proportion of patients with adverse events, and frequency and grade of each AE (assessment of safety and tolerability to G-MTF) | During treatment and after the follow up peridod (total of 4 month)
  The number and percentage of patients experiencing each adverse event (AE), as well as the frequency and grade of each AE, will be assessed. Throughout the treatment and follow-up period, the presence or absence of AEs at both local and systemic levels will be monitored in each of the five patients included in the G-MTF groups (G-MTF 0.5%, 1.0%, and 1.5%). Each AE will be graded on a scale from 0 to 3:
  * 0 indicates absence of the AE;
  * 1 denotes mild severity (present but not requiring treatment);
  * 2 indicates moderate severity (present and requiring specific treatment);
  * 3 signifies severe severity (present with such intensity that antileishmania therapy must be discontinued).
  These grades follow the Common Terminology Criteria for Adverse Events (CTCAE).

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Blanco, PhD, Study Chair — Universidad Industrial de Santander
Locations (1):
- Calle 158 No. 20-95 Cañaveral, Floridablanca, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neira LF, Mantilla JC, Escobar P. Monitoring cutaneous leishmaniasis lesions in mice undergoing topical miltefosine treatment. Sci Pharm. 2023; 91(4):54. https://doi.org/10.3390/scipharm91040054
- [Background] Neira LFb., Peña DP., Vera AM., Mantilla JC., Escobar P. Leishmaniasis cutánea inducida por especies de Leishmania Viannia en ratones BALB/c y eficacia de un tratamiento tópico. Rev Univ Ind Santander. Salud. 2019 Mar;51(1):33-42.doi.org/10.18273/ revsal.v51n1-2019004
- [Background] Neira LF, Mantilla JC, Escobar P. Anti-leishmanial activity of a topical miltefosine gel in experimental models of New World cutaneous leishmaniasis. J Antimicrob Chemother. 2019 Jun 1;74(6):1634-1641. doi: 10.1093/jac/dkz049. PMID 30815688
- [Background] Escobar P, Yardley V, Croft SL. Activities of hexadecylphosphocholine (miltefosine), AmBisome, and sodium stibogluconate (Pentostam) against Leishmania donovani in immunodeficient scid mice. Antimicrob Agents Chemother. 2001 Jun;45(6):1872-5. doi: 10.1128/AAC.45.6.1872-1875.2001. PMID 11353640
- [Background] Castro MD, Gomez MA, Kip AE, Cossio A, Ortiz E, Navas A, Dorlo TP, Saravia NG. Pharmacokinetics of Miltefosine in Children and Adults with Cutaneous Leishmaniasis. Antimicrob Agents Chemother. 2017 Feb 23;61(3):e02198-16. doi: 10.1128/AAC.02198-16. Print 2017 Mar. PMID 27956421
- [Background] Blum J, Lockwood DN, Visser L, Harms G, Bailey MS, Caumes E, Clerinx J, van Thiel PP, Morizot G, Hatz C, Buffet P. Local or systemic treatment for New World cutaneous leishmaniasis? Re-evaluating the evidence for the risk of mucosal leishmaniasis. Int Health. 2012 Sep;4(3):153-63. doi: 10.1016/j.inhe.2012.06.004. PMID 24029394
- [Background] Aronson N, Herwaldt BL, Libman M, Pearson R, Lopez-Velez R, Weina P, Carvalho E, Ephros M, Jeronimo S, Magill A. Diagnosis and Treatment of Leishmaniasis: Clinical Practice Guidelines by the Infectious Diseases Society of America (IDSA) and the American Society of Tropical Medicine and Hygiene (ASTMH). Am J Trop Med Hyg. 2017 Jan 11;96(1):24-45. doi: 10.4269/ajtmh.16-84256. Epub 2016 Dec 7. No abstract available. PMID 27927991
- [Background] Andrade HM, Toledo VP, Pinheiro MB, Guimaraes TM, Oliveira NC, Castro JA, Silva RN, Amorim AC, Brandao RM, Yoko M, Silva AS, Dumont K, Ribeiro ML Jr, Bartchewsky W, Monte SJ. Evaluation of miltefosine for the treatment of dogs naturally infected with L. infantum (=L. chagasi) in Brazil. Vet Parasitol. 2011 Sep 27;181(2-4):83-90. doi: 10.1016/j.vetpar.2011.05.009. Epub 2011 May 14. PMID 21641721